CLINICAL TRIAL: NCT06031948
Title: Personalized Brain Functional Sectors (pBFS) Guided Noninvasive Neuromodulation Treatment for Pre-school Children With Autism Spectrum Disorder (ASD): a Single-center, Double-blinded, Sham-Controlled, Randomized Clinical Trial Study
Brief Title: pBFS-guided Noninvasive Neuromodulation for Pre-school Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changping Laboratory (Other)
Collaborators: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLASD2023HNC50
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Autism Spectrum Disorder
Keywords: TMS; ASD; fMRI; personalized medicine
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DLPFC group (Experimental): Active iTBS will be delivered to the left DLPFC.
  Interventions: Device: active iTBS
- DMPFC group (Experimental): Active iTBS will be delivered to the left DMPFC.
  Interventions: Device: active iTBS
- Sham to DLPFC group (Sham Comparator): Sham iTBS will be delivered to the left DLPFC.
  Interventions: Device: sham iTBS
- Sham to DMPFC group (Sham Comparator): Sham iTBS will be delivered to the left DMPFC.
  Interventions: Device: sham iTBS

INTERVENTIONS:
Device: active iTBS — Each participant will receive 1800 pulse active iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 8 weeks.
  Arms: DLPFC group
Device: active iTBS — Each participant will receive 1800 pulse active iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 8 weeks.
  Arms: DMPFC group
Device: sham iTBS — Each participant will receive 1800 pulse sham iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 8 weeks.
  Arms: Sham to DLPFC group
Device: sham iTBS — Each participant will receive 1800 pulse sham iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 8 weeks.
  Arms: Sham to DMPFC group

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy and safeness of the pBFS-guided rTMS intervention for core symptom relief in pre-school children with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
Autism spectrum disorder is a neurodevelopmental disorder, begins early in life. Using the personalized brain functional sectors (pBFS) technology, investigators could precisely identify individualized brain function networks based on the functional MRI scan. For each participant, two personalised TMS intervention targets will be chosen by blinded researcher. One executive function network target is located in the dorsal lateral prefrontal cortex (DLPFC) , and the other social function network target is located in the dorsal medial prefrontal cortex (DMPFC).

The participants will be equally randomized to the following four groups, active iTBS to the left DMPFC or the left DLPFC, and sham iTBS to either the left DMPFC or left DLPFC at a ratio of 2:2:1:1. Later analyses will combine the two sham groups as one control group. Each participant will receive 1800 pulse active or sham iTBS (100% RMT) in each session, 3 sessions daily, 5 days per week for 8 weeks, as well as background behavioral training between iTBS sessions. Pre-and post-treatment functional MRI data will be collected under sedation.

ELIGIBILITY:
Inclusion Criteria:

* 2.5-6 years old
* Have the diagnosis of autism spectrum disorder
* ADOS-2 score is higher than the ASD cut-offs
* Capacity to follow the study procedures, including fMRI scan under sedation, assessment, and rehabilitation training
* Participant's parents or other legal guardians give informed consent

Exclusion Criteria:

* Current or history of psychotic disorders, such as schizophrenia, schizoaffective disorder, bipolar disorder
* Severe self-injury or suicidal behavior presented in the last 1 year
* Severe visual, auditory, or motor disability that interferes with any study procedure
* Current, history or family history of epilepsy
* Known severe physical diseases, such as congenital heart defect, traumatic brain injury
* Metal implantations, which are contradicted by MRI or TMS, such as artificial cardiac pacemakers, stents, cochlear implants
* Received TMS, tCS, FUS, or other neuromodulation treatment in the last 3 months
* Currently participating in other clinical trials

Ages: 30 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
ADOS-2 SA change | Pre-treatment (baseline), immediately post-treatment
  The social affect (SA) dimension score change of autism diagnostic observation scale, 2nd edition (ADOS-2) from baseline. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
ADOS-2 total score change | Pre-treatment (baseline), immediately post-treatment
  The total score change of autism diagnostic observation scale, 2nd edition (ADOS-2) from baseline. Higher scores mean a worse outcome.
CBCL score change | Pre-treatment (baseline), immediately post-treatment
  Score change of the child behavior checklist (CBCL) from baseline. Higher scores mean a worse outcome.

OTHER OUTCOMES:
SCQ score change | Pre-treatment (baseline), immediately post-treatment
  Score change of the Social Communication Questionnaire (SCQ) from baseline. Higher scores mean a worse outcome.
SRS-2 score change | Pre-treatment (baseline), immediately post-treatment
  Score change of the Social Responsiveness Scale, 2nd edition (SRS-2) from baseline. Higher scores mean a worse outcome.
RBS-R score change | Pre-treatment (baseline), immediately post-treatment
  Score change of the Repetitive Behavior Scale-Revised (RBS-R) from baseline. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory